CLINICAL TRIAL: NCT06779240
Title: Non-specific Low Back Pain and Low Back Pain Secondary to Scoliosis: is It Possible to Differentiate Them Through Quality of Life Questionnaires?
Brief Title: Distinguishing Non-Specific Low Back Pain from Scoliosis-Related Pain Via Quality of Life Questionnaires
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: LBP-Scoliosis
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Scoliosis; Degenerative Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Scoliosis patients: Patients with a diagnosis of idiopathic scoliosis or degenerative scoliosis
  Interventions: Other: Quality of life questionnaires
- Non specific LBP: Patients with non specific low back pain
  Interventions: Other: Quality of life questionnaires

INTERVENTIONS:
Other: Quality of life questionnaires — The clinical protocols at our institute involve the regular and continuous evaluation of the quality of life in patients undergoing treatment and monitoring for scoliosis and other vertebral deformities. To this end, the SRS-22 (Scoliosis Research Society) questionnaire and the ODI (Oswestry Disability Index) questionnaire are employed, along with other measures such as the COMI (Core Outcome Measure Index) and ISYQoL (Italian Spine Youth Quality of Life) and administrated to every patients

SUMMARY:
Vertebral deformities, such as scoliosis, can have a significant impact on the physical and psychological health of patients. Over time, specific tools have been developed to investigate the extent of this impact; the SRS-22 (Scoliosis Research Society) questionnaire is the most commonly used instrument for assessing quality of life (QoL) in patients with idiopathic scoliosis. The Oswestry Disability Index (ODI), on the other hand, was developed to evaluate the quality of life in adult patients with chronic non-specific low back pain.

The clinical protocols at our institute involve the regular and continuous evaluation of the quality of life in patients undergoing treatment and monitoring for scoliosis and other vertebral deformities. To this end, the SRS-22 questionnaire and the ODI questionnaire are employed, along with other measures such as the COMI (Core Outcome Measure Index) and ISYQoL (Italian Spine Youth Quality of Life).

The aim of this study is to compare the properties of the ODI with those of the SRS-22 questionnaire in adults, by analyzing differences between individuals with non-specific low back pain and those with scoliosis. The secondary objective involves a sub-analysis based on the severity of scoliosis, dividing curves into major (30° Cobb or higher) and minor (below 30° Cobb). Finally, if sufficient data are available, the study will also evaluate other commonly used questionnaires (COMI and ISYQoL).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of idiopathic or degenerative scoliosis with a curve >10° Cobb and
* low back pain
* Diagnosis of non-specific low back pain

Exclusion Criteria:

* Previous spinal surgery
* Significant past illnesses, surgeries, or trauma
* Secondary scoliosis
* Other deformities such as spondylolisthesis and spinal canal stenosis
* Incomplete ODI and SRS-22 data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with LBP or scoliosis accessing a tertiary referral outpatient clinic specialized in the conservative treatment of spinal deformities
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaires comparison | through study completion, an average of 1 year
  compare the properties of the Oswestry Disability Index (ODI) with those of the SRS-22 questionnaire in adults, specifically by analyzing differences between individuals with non-specific low back pain and those with scoliosis.
  This comparison focuses on determining the effectiveness and applicability of these tools in assessing quality of life (QoL) in these two distinct patient populations.

CONTACTS AND LOCATIONS:
Locations (1):
- ISICO, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided